CLINICAL TRIAL: NCT06850194
Title: Evaluating the Efficacy of Vertical Ramus Osteotomy With Iliac Graft Versus Bilateral Sagittal Split Osteotomy for the Correction of Mandibular Deficiency in Skeletal Class II Cases Management. A Randomized Controlled Trial
Brief Title: Vertical Ramus Osteotomy With Iliac Graft Versus Sagittal Split Osteotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor oral and maxillofacial surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Mandibular Deficiency
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Sagittal Split Osteotomy Group (Active Comparator)
  Interventions: Procedure: bilateral sagittal splitting osteotomy
- vertical ramus osteotomy with iliac graft group (Experimental)
  Interventions: Procedure: vertical ramus osteotomy with iliac graft

INTERVENTIONS:
Procedure: vertical ramus osteotomy with iliac graft — in the VRO group all patient will undergo vertical ramus osteotomy surgery with iliac graft to correct the sever mandibular defficiency
  Arms: vertical ramus osteotomy with iliac graft group
Procedure: bilateral sagittal splitting osteotomy — all patients in this group will undergo to bilateral sagittal split osteotomy to correct the sever mandibular deficiency
  Arms: Bilateral Sagittal Split Osteotomy Group

SUMMARY:
* Patients will be collected from faculty of dentistry
* bilateral vertical ramus osteotomy (VRO )with iliac graft group (group I):- 10 patients will be treated via VRO and iliac crest or
* bilateral sagital spilt osteotomy (BSSO) group (group II):- 10 patients will be treated via BSSO
* All patients will be studied by comprehensive clinical oral and maxillofacial examination and lateral cephalometric radiographic analyses, within 1 week before the surgery (T0), immediately after the surgery (T1), and 6 months after surgery (T2).
* All lateral cephalometric radiographs and clinical photographs must be standardized for all cases.
* After pre-surgical orthodontic treatment , a lateral cephalograph Will be obtained for planning the surgical movement of both jaws
* Surgical models and surgical stent will be fabricated.
* All surgical procedures will be performed under nasal intubation and general anesthesia to surgically reposition the maxilla in standard LeFort I setback fosteotomy; the BSSO group will be underwent BSSO, and VRO group will be underwent VRO
* The bony segments will be fixed in the new position with the use of custom made plates (specific for each patient )

ELIGIBILITY:
Inclusion Criteria:

* patients with age above 18 years old suffered from skeletal class II with severe mandibular deficiency

Exclusion Criteria:

* patients with chin deviation,
* severe temporomandibular joint (TMJ) symptoms.
* Sever periodontal disease
* pregnancy,
* previous mandibular surgery,
* inability to follow-up for the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
skeletal stability | 6 months
  Skeletal stability will be assessed by lateral cephalometric x-ray. It will be done pre operatively, immediate postoperative, and 6 months later

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suief University, Beni-seuf, Egypt, Egypt